CLINICAL TRIAL: NCT02454738
Title: Ultralow Dose Computed Tomography in Close Contacts at High Risk for Developing Multidrug- or Extensively Drug-resistant Tuberculosis: A Pilot Study
Brief Title: Ultralow Dose Computed Tomography in High-risk Drug-resistant Tuberculosis Contacts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Mo Goo, Professor, Department of Radiology, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUHchestradiology-001
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Latent Tuberculosis
Keywords: pulmonary tuberculosis; chest; ultralow dose computed tomography
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chest CT scan (Experimental): Two follow-up ultralow dose chest CT scans will be taken 3 months and 1 year after the initial ultralow dose chest CT scan in close contact at high risk for developing multidrug- or extensively drug-resistant tuberculosis.
  Interventions: Radiation: Ultralow dose chest CT scan

INTERVENTIONS:
Radiation: Ultralow dose chest CT scan — Ultralow-dose chest CT scan is performed using a 64-row multidetector CT system (Discovery CT750HD; GE Healthcare, Waukesha, WI) with 1.25-mm-thick axial slices at less than 1 mSv (volume computed tomography dose index: 0.39 milligray).

SUMMARY:
To evaluate CT abnormalities in the lung parenchyma in close contacts at high risk for developing multidrug- or extensively drug-resistant Tb by using a follow-up ultralow dose CT scan.

DETAILED DESCRIPTION:
Multidrug- or extensively resistant tuberculosis tuberculosis is a major public health threat worldwide and the global burden of drug-resistant tuberculosis is increasing. Drug-resistant tuberculosis is associated with long period and high costs for treatment, high rates of default, treatment failure and death.

Drug-resistant tuberculosis should be diagnosed rapidly so as to reduce potential transmission. In the United States, at least one-fifths cases of multidrug-resistant tuberculosis can be linked to transmission. Close contacts to drug-resistant tuberculosis are at high risk for being transmitted and developing drug-resistant tuberculosis. There are two options suggested for close contacts to drug-resistant tuberculosis: preventive therapy and close observation. But both strategies are lack of sufficient evidence.

Ultralow chest CT scan may be an alternative for early identification and risk stratification of developing active tuberculosis in close contacts to drug-resistant tuberculosis with minimal radiation exposure similar to that of chest x-ray.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who had household contact with or who had worked in the same rooms as patients with smear-positive, culture-proven multidrug-or extensively drug-resistant pulmonary tuberculosis for longer than 8 hours per day
* Older than 20 years

Exclusion Criteria:

* Pregnant women
* Individuals with abnormality on chest x-ray suspected of active tuberculosis

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Interval change of CT abnormalities potentially suggesting active tuberculosis in the lung parenchyma during the follow-up. | 3 months and 1 year after the initial CT scanning

CONTACTS AND LOCATIONS:
Overall Officials: Jin Mo Goo, M.D., Principal Investigator — Department of Radiology, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lee SC, Yoon SH, Goo JM, Yim JJ, Kim CK. Submillisievert Computed Tomography of the Chest in Contact Investigation for Drug-Resistant Tuberculosis. J Korean Med Sci. 2017 Nov;32(11):1779-1783. doi: 10.3346/jkms.2017.32.11.1779. PMID 28960029